CLINICAL TRIAL: NCT06519435
Title: Non-invasive Venous Air Plethysmography Assessment of Venous Hemodynamics in Patients Suspected Deep Venous Obstruction Used in Conjunction With Intermittent Pneumatic Compression.
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Damon E. Houghton, Physician, Vascular Medicine, Mayo Clinic
Other Study IDs: 23-012242
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Mayo Dopplex ABIlity — Device used to measure lower extremity venous hemodynamic pressure
Device: Intermittent Pneumatic Compression (IPC) — Device used to measure lower extremity venous hemodynamic pressure

SUMMARY:
The purpose of this research is to measure changes in venous blood flow with an air-filled bladder under an intermittent pneumatic compression device cuff (used to prevent deep venous thrombosis) or venous diagnostic device cuff (used to detect deep venous thrombosis). The devices being used in the study are investigational and not FDA-cleared.

ELIGIBILITY:
Inclusion Criteria:

* Venous ultrasound study to evaluate for lower extremity DVT unilateral and/or bilateral within previous 72 hours.

Exclusion Criteria:

* Patients with inaccessible target limb (ultrasound limb) due to bandages (wound, burn, lesion, etc) or cast.
* Patients with leg trauma, fracture, above or below knee amputation, or other condition in which compressing on the calf is medically inappropriate or not possible.
* Patients unable to provide informed written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with venous ultrasound evaluation performed to rule out deep vein thrombosis
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Mayo Dopplex ABllity device Venous hemodynamic pressure | Baseline
  Venous hemodynamic pressure to be measured from both the recumbent and sitting positions using the Mayo Dopplex ABllity device. Measured as mmHg.
Intermittent Pneumatic Compression device Venous hemodynamic pressure | Baseline
  Venous hemodynamic pressure to be measured from both the recumbent and sitting positions using the IPC device. Measured as mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Damon Houghton, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No